CLINICAL TRIAL: NCT04263272
Title: Circuit Training Program Tom Improve Endocrine-Metabolic Function in Persons With Spinal Cord Injury
Brief Title: Circuit Training Program for Persons With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Dalton Wolfe, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 113642
Record Dates: First submitted 2019-12-05; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Injuries
Keywords: Endocrine-Metabolic health; Cardio-Metabolic health
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upper Body Exercise (Experimental): Seated upper body circuit training program for 16-weeks. Frequency - 1 to 3 one-hour sessions per week.
  Interventions: Other: Upper Body Circuit Training Program

INTERVENTIONS:
Other: Upper Body Circuit Training Program — 16 week seated upper body exercise for persons with Spinal Cord Injuries. Participants will attend 2-3 exercise sessions a week, sessions have a mix of SCI community members and inpatients.

SUMMARY:
This initiative represents development and pilot testing of a circuit training exercise program for persons with spinal cord injury (SCI) to be implemented within a rehabilitation centre. The program will integrate members of the community who are > 18 months post-injury with those currently participating in SCI rehabilitation as inpatient.

DETAILED DESCRIPTION:
This initiative represents development and pilot testing of a 16 week circuit training exercise program for persons with spinal cord injury (SCI) to be implemented within a rehabilitation centre (Parkwood Institute, London, ON). The primary purpose of this trial is one of feasibility - i.e., testing out several aspects of the trial for the purposes of determining what features of the exercise intervention and the various outcome measurements might be a part of subsequent trials. In addition, a subset of this data will serve as preliminary comparison information for Dr. Dany Gagnon's study at the University of Montreal. In this way, this is not a true multi-centre trial in that we are not conducting an identical protocol to a study he is conducting. Rather, we are using some of the same outcome measures and an exercise intervention that has some similar parameters to one that he is implementing in Montreal - with a view to providing a preliminary comparison of outcomes of a subset of participants in our study so as to inform the development of future studies. For this reason, the group of community-dwelling persons with SCI will have more cardio-metabolic outcome measurements taken, as they represent the primary group of interest to Dr. Gagnon.

Overall, the program will integrate members of the community who are > 18 months post-injury (n=8) with those currently participating in SCI rehabilitation as inpatients (n=8). Outcomes will be collected to test the effects of the program on an array of cardio-metabolic measures in those participants with chronic SCI, as well as the feasibility of the program for all participants (N=16). Note: although a participant can decline to continue participation at any time, it is likely that many inpatient participants will choose to not continue participation if this proves logistically difficult (if they move back to their home community away from London).

ELIGIBILITY:
Inclusion Criteria:

Community:

* Chronic traumatic or non-traumatic SCI between level C6 and T10 >18 months post injury
* manual wheelchair as the primary mode of mobility
* no existing conditions that would make it unsafe to participate in an exercise program (e.g., fractures).
* Ability to understand and communicate in English.
* 18 years or older.

Inpatients:

* Chronic traumatic or non-traumatic SCI between level C6 and T10
* manual wheelchair as primary mode of mobility
* no existing conditions that would make it unsafe to participate in an exercise program (e.g., fractures).
* Ability to understand and communicate in English.
* 18 years or older.

Exclusion Criteria:

* Power wheelchair users (Non manual wheelchairs)
* Have an existing condition that would make it unsafe to participate in an exercise program (e.g., fracture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility survey | After Study Completion (16 weeks)
  Feasibility question options range from -3 to +3 on a likert scale, higher scores indicated a greater level of feasibility.
Injury Characteristics Survey | Baseline
  Date of injury (DD/MM/YYYY)
Injury Characteristics Survey | Baseline
  Diagnosis - Traumatic SCI or Non-Traumatic SCI
Injury Characteristics Survey | Baseline
  Classification of SCI using the AIS (ASIA Impairment Scale) - A, B, C, D or E
Injury Characteristics Survey | Baseline
  Neurological Level or Injury (NLI)
Change in Spinal Cord Injury Independence Measure - Mobility | Baseline and 16 weeks
  Assessment of degree to which participant can independently preform mobility tasks, such as transfers, and the ue of mobility aids.
Change in Upper and Lower Extremity Strength by a manual muscle test (MMT) | Baseline and 16 weeks
  Assessment of joint (Shoulder, elbow, wrist, hip, knee and ankle) muscle strength using a Manual muscle test.
Change in Upper and Lower Extremity Range of Motion | Baseline and 16 weeks
  Assessment of joint range of motion in the upper and lower extremities (Shoulder, elbow, wrist, hip, knee and ankle)
Change in Spasticity in upper and lower extremities using the Modified Ashworth Scale | Baseline and 16 weeks
  Assessment of muscle tone through range of motion, on a scale of 0-4 (0= no increase in muscle tone; 4 = rigidity in flexion or extension)
Change in Maximal Safe Wheel chair speed measured using the Propulsion Speed Test | Baseline and 16 weeks
  20 meter straight line wheel chair speed test. 3 trails were be preformed at a comfortable speed and 3 trials will be preformed at a maximal but safe speed.
Change in Ability to safety navigate wheel chair using the Slalmon Speed test | Baseline and 16 weeks
  Objective is to weave between a set of cones without touching them as fast as safely possible. 3 attempts will be given.
Demographics and Lifestyle Questionnaires | Baseline
  Age in years
Demographics and Lifestyle Questionnaires | Baseline
  Gender (Women, Man or Other)
Demographics and Lifestyle Questionnaires | Baseline
  Marital Status
Demographics and Lifestyle Questionnaires | Baseline
  Ethnicity
Demographics and Lifestyle Questionnaires | Baseline
  Highest Education Level completed
Demographics and Lifestyle Questionnaires | Baseline
  Currently Employment situation
Demographics and Lifestyle Questionnaires | Baseline
  Family income ($ in last year)
Demographics and Lifestyle Questionnaires | Baseline
  List of Medical/health problems
Demographics and Lifestyle Questionnaires | Baseline
  Smoking levels (yes/no and how many years)
Demographics and Lifestyle Questionnaires | Baseline
  Cannabis Use (yes/no, frequency, types of products)
Demographics and Lifestyle Questionnaires | Baseline
  Vaping (Yes/no, frequency)
Demographics and Lifestyle Questionnaires | Baseline
  Alcohol consumption (frequency and beverages consumed when drinking)
Demographics and Lifestyle Questionnaires | Baseline
  Physical Activity levels (minutes/week)
Change in Medications | Baseline and 16 weeks
  List of medication and supplements currently being taken.
Change in Experienced Pain | Baseline and 16 weeks
  The international Spinal Cord Injury Pain Data Set will be used to evaluate the presence and severity of pain. Description of 3 main pain concerns and there intensity. Intensity ranges from 0 = no pain to 10 = worst possible pain.
Change in Wheel Chair skills ability using the Wheel Chair skills Test Questionnaire | Baseline and 16 weeks
  Questionnaire assesses the ability and confidence in preforming numerous wheel chair skills (ex: turning the wheelchair around a small space) Questions answers include 'No' 'partially' 'yes' 'very well'.
Change in Well Being measured by the General Wellbeing Index | Baseline and 16 weeks
  Assessment of emotional wellbeing, on a scale of 0-5.
Change in Quality of life and health measured by the WHOQOL-BREF | Baseline and 16 weeks
  Self reported questionnaire assessing quality of life (physical, social, environment and psychological health) on a scale of 1 - 4 (1=poor/not al all; 5= very good/extreme amount)
Change in aerobic capacity (VO2max) measured by 6-min wheelchair propulsion test | Baseline and 16 weeks
  Objective is to get the largest total distance. Pylons are placed 25meters apart, participants starts in the middle go around the first cone to the let return to the middle and make a full stop, then continue to the right of second cone, go around it and back to the middle, making a figure 8. Continue that pattern for 6 minutes.
Blood Test | Baseline and 16 weeks
  Measurement of metabolic profile (ex: glucose, insulin, triglyceride)
Blood Test | Baseline and 16 weeks
  Measurement of bone markers (ex: osteocalcin)
Change in Body composition measured by DEXA (Dual energy x-ray absorptiometry) | Baseline and 16 weeks
  Measurement of bone mineral density of the full body (reported using a T score)
Change in Body composition measured by DEXA (Dual energy x-ray absorptiometry) | Baseline and 16 weeks
  Measurement of bone mineral density of the femoral head (reported using a T score)
Change in Body composition measured by DEXA (Dual energy x-ray absorptiometry) | Baseline and 16 weeks
  Measurement of bone mineral density of the lumbar spine (reported using a T score)

CONTACTS AND LOCATIONS:
Overall Officials: Dalton Wolfe, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's